CLINICAL TRIAL: NCT06461702
Title: Clinical Exploration Trial of YOLT-101 in the Treatment of Familial Hypercholesterolemia (FH)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FH-YOLT-101-1
Record Dates: First submitted 2024-04-16; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-04

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YOLT-101 (Experimental)
  Interventions: Drug: YOLT-101

INTERVENTIONS:
Drug: YOLT-101 — The IP is administered intravenously at the predetermined dose.

SUMMARY:
This study is a single arm, open, single dose escalation trial aimed at evaluating the safety and tolerability of YOLT-101 administration in patients with familial hypercholesterolemia; Determination of YOLT-101 OBD; Preliminary evaluation of the effects of single administration of YOLT-101 on plasma lipid and lipoprotein levels.

Note: OBD is defined as the dosage at which plasma PCSK9 protein levels decrease between 60% and 95% from baseline on the 28th day after YOLT-101 administration. OBD ≤ Maximum Tolerable Dose (MTD).

DETAILED DESCRIPTION:
In this study, the longest screening period for the main study was 42 days, the treatment day was Day 1 (D1), and the safe follow-up period was up to 52 weeks after medication. In the main study, when OBD occurs, additional subjects will be added to the dose group (specific number of cases will be negotiated between the cooperating organization and investigators) for further validation. In addition, subjects in the first dose group can voluntarily receive a second drug administration of OBD level.

After the completion of the main study, participants will undergo long-term follow-up. According to the Technical Guidelines for Long term Follow up Clinical Research of Gene Therapy Products (Trial) released by CDE, a long-term follow-up until 15 years after the medicine administration is required .

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged ≥ 18 years and ≤ 65 years (including boundary values) who signed informed consent.
2. Meets the diagnostic criteria for familial hypercholesterolemia. When screening, there are mutations in the PCSK9 and/or ApoB and/or LDLR genes.

4. When screening, the weight should be ≥ 40kg, and the body mass index (BMI) should be between 18-30 kg/m2 (including boundary values).

5. During screening, subjects must meet the following laboratory standards: 5.1 Blood routine: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 100 × 109/L, hemoglobin count (HGB) ≥ 90 g/dL; 5.2 Liver function: aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) < 2.0 × ULN, total bilirubin (TBIL) ≤ 1.5 × ULN; 5.3 Renal function: Serum creatinine (Cr) ≤ 1.5 × ULN, and glomerular filtration rate (GFR)>60mL/min * 1.73m2; 5.4 Coagulation function: prothrombin time (PT), activated partial thromboplastin time (APTT), international standardized ratio (INR)<1.5 x ULN; 5.5 Low density lipoprotein cholesterol (LDL-C) ≥ 4.21mmol/L, and fasting triglycerides<5.6mmol/L.

6. The subjects and their partners must take effective contraceptive measures during the participation in this study until 6 months after the end of the main study.

7. The subject must agree not to accept other lipid-lowering drugs for at least 28 days after receiving the investigational drug.

8. Voluntarily sign informed consent.

Exclusion Criteria:

1. Those who have used any prescription drugs that affect blood lipid metabolism within at least 14 days before receiving the study drug (or within 7 half lives of the drug, whichever is longer, applicable to small molecule/small nuclear acid drugs) or within 3 months (applicable to biological agents such as PCSK9 inhibitors), or who have used any over-the-counter drugs that affect blood lipid metabolism within at least 14 days before receiving the study drug (such as Chinese medicine/traditional Chinese patent medicines and simple preparations, vitamins, fish oil (>1000mg/day), drugs containing red koji rice or health products, etc.), (Exception of those who have received stable non-cyclical hormone replacement therapy for more than 8 weeks and agree not to change the hormone treatment more than 28 days after the study drug administration); individuals who have participated in clinical studies of other lipid-lowering drugs and have accepted the investigational drugs within 6 months before the screening period.
2. Poorly controlled hypertensive patients who have receive conventional treatments (systolic blood pressure (SBP) ≥ 160mmHg and/or diastolic blood pressure (DBP) ≥ 100mmHg).
3. Poorly controlled diabetes patients (glycosylated hemoglobin>8.5%).
4. Individuals who are allergic to drugs or mRNA vaccine components contained in lipid nanoparticles (LNPs), or have experienced adverse reactions to LNP drug therapy, such as:

   4.1 After receiving LNP drug treatment, ALT or AST>3.0 × ULN; 4.2 After receiving LNP drug treatment, INR>1.5 or APTT/d-dimer>1.5 × ULN; 4.3 Any infusion response that requires clinical intervention, slows down infusion rate, or stops LNP drugs treatment; 4.4 Any other adverse reactions that researchers believe are related to the treatment of LNP drugs.
5. Within three months before the screening, individuals who smoke more than 5 cigarettes per day or consume an equal amount of nicotine or nicotine substitutes.
6. Individuals with a history of alcohol abuse [consuming more than 14 units of alcohol per week (1 unit ≈ 360mL of beer or 45mL of 40% liquor or 150mL of wine)] within 3 months before the screening; Individuals positive for alcohol breath test during the screening or admission.
7. Grade III-IV heart failure defined by the New York Heart Association (NYHA), or left ventricular ejection fraction<50%, or prolonged QTc interval (>470ms in females and>450ms in males) found during the screening.
8. Suffering poorly controlled severe arrhythmia , such as recurrent and highly symptomatic ventricular tachycardia with poorly drug controlled, atrial fibrillation with rapid ventricular reaction, or supraventricular tachycardia within three months before the screening.
9. Myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass grafting, severe deep vein thrombosis or pulmonary embolism within three months before the screening; Cerebrovascular accidents occurring within 6 months before the screening or planning for cardiac surgery or revascularization during the main study period.
10. Suffering from diseases that have a significant impact on blood lipid levels and cannot be controlled, such as nephrotic syndrome, severe liver disease, Cushing's syndrome, thyroid dysfunction, etc. (Individuals with hypothyroidism who have undergone stable thyroid replacement therapy for ≥ 28 days before screening, have normal TSH testing, and agree to maintain the dose of thyroid replacement drugs unchanged during the study can be considered to be enrolled).
11. Individuals who have donated more than 500 mL of blood within three months before screening.
12. Those who are unable or unwilling to accept the medication treatment required before the investigational treatment.
13. Patients who underwent antithrombotic treatment (such as warfarin, dabigatran, and apixaban) within 14 days prior to enrollment.
14. Those who are prone to bleeding or have a history of coagulation disorders (such as cirrhosis, malignant hematological diseases, antiphospholipid antibody syndrome);
15. Patients with an expected survival period of less than 2 years.
16. Individuals who are known or suspected to have systemic viral, parasitic, or fungal infections, or are expected to receive antibiotic treatment within 14 days after screening.
17. Hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody positive during the screening.
18. Individuals who have received liver, heart, or other solid organ transplantation, bone marrow transplantation within one year before the screening, or having a transplantation plan during the clinical trial.
19. Individuals with a history of malignant tumors within 5 years before the screening (excluding curative skin basal cell carcinoma, skin squamous cell carcinoma, cervical carcinoma in situ, low-grade prostate carcinoma in situ, and curative thyroid basal carcinoma in situ).
20. Individuals with a history of drug use within three years before the screening.
21. Pregnant or lactating women.
22. Patients with other systemic diseases such as the blood system, digestive system, or central nervous system (including cerebrovascular diseases and degenerative diseases) that the researchers believe will interfere with the evaluation or limit the participation in the trial.
23. Severe mental diseases that researchers believe which cannot be fully controlled by the medication treatment.
24. Those who are unwilling to follow the research procedures or are unwilling to fully cooperate.
25. Other situations that researchers believe not suitable to participate in the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
safety evaluation of YOLT-101 | through week 52
  The safety of YOLT-101 evaluated by the proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs)

SECONDARY OUTCOMES:
pharmacokinetics of YOLT-101 | through Day 28
  The Peak Plasma Concentration (Cmax) of YOLT-101. 0.5 predose,0.5,1,1.5,2,4,6,8,12,24,48,72,144,312 hours
pharmacodynamics | through week 52
  The effect of YOLT-101 on serum levels of LDL-C
pharmacodynamics | through week 52
  The effect of YOLT-101 on plasma levels of PCSK9
pharmacokinetics of YOLT-101 | through Day 28
  Area under the plasma concentration versus time curve (AUC). 0.5 predose,0.5,1,1.5,2,4,6,8,12,24,48,72,144,312 hours
pharmacokinetics of YOLT-101 | through Day 28
  Tmax
pharmacokinetics of YOLT-101 | through Day 28
  T1/2

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui, China

IPD SHARING:
Plan to Share IPD: No